CLINICAL TRIAL: NCT02507232
Title: A Multicenter, Open-Label, Randomized Study of NovoTTF-200A Alone and Combined With Temozolomide in Patients With Low-Grade Gliomas
Brief Title: Study of NovoTTF-200A Alone and With Temozolomide in Patients With Low-Grade Gliomas
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Santosh Kesari (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Santosh Kesari, Associate Professor, Saint John's Cancer Institute
Organization: Saint John's Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JWCI-16-1101
Record Dates: First submitted 2015-07-21; First posted 2015-07-23 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Glioma
Keywords: glioma; temozolomide; brain; NovoTTF-200A; cancer; low-grade glioma
MeSH Terms: conditions — Glioma; Neoplasms | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm A (Active Comparator): NovoTTF-200A
  Interventions: Device: NovoTTF-200A
- Arm B (Active Comparator): NovoTTF-200A + Temozolomide 50 mg/m2 daily (oral)
  Interventions: Device: NovoTTF-200A; Drug: Temozolomide

INTERVENTIONS:
Device: NovoTTF-200A — 12 cycles
Drug: Temozolomide — 50 mg/m2/day rounded to the nearest 5 mg. One cycle is 28 days and will be given for 12 cycles
  Other Names: Temodar
  Arms: Arm B

SUMMARY:
The purpose of this study is to test the effectiveness and safety of the NovoTTF-200A device in patients with low-grade glioma when it's used by itself or used together with temozolomide. Researchers would also like to know whether the use of NovoTTF-200A, with or without temozolomide, is associated with fewer negative side effects on mental function that may be seen with other currently used treatment options.

DETAILED DESCRIPTION:
Approximately 2,000 to 3,000 low-grade gliomas (LGGs) are diagnosed in adults each year in the United States. Based on a variety of prognostic factors the median overall survival ranges from 3 to 9 years.

NovoTTF-200A is a device that produces alternating electrical fields within the human body that disrupt cell division. These very low intensity intermediate frequency electric fields (TTFields) impair the growth of tumor cells through the arrest of cell division and inducing apoptosis.

Although FDA approved for the treatment of recurrent or progressive glioblastoma, further investigation of NovoTTF-200A is warranted, in the setting of low-grade glioma where it has the potential to stunt tumor growth without significant toxicity. NovoTTF-200A has also been shown to be safe combined with adjuvant 5-day temozolomide regimen in newly diagnosed glioblastoma in an ongoing clinical trial. Given the low proliferative index in low-grade gliomas, combining NovoTTF-200A with metronomic chemotherapy may be more effective.

This is a randomized, 2-arm, open label study of NovoTTF-200A alone or combined with daily temozolomide for the treatment of patients with newly diagnosed low-grade gliomas.

Patients will be randomized 1:1 to one of two arms for a total of 22 patients (11 per arm). Arm A will receive NovoTTF-200A only and Arm B will receive NovoTTF-200A and low-dose (50 mg/m2) daily temozolomide regimen.

All patients providing informed consent will be screened for eligibility. Baseline assessments will include vital signs, physical exam, blood hematology and chemistries, Karnofsky Performance Status (KPS) evaluation, Quality of Life (QOL) assessment using the Functional Assessment of Cancer Therapy-Brain (FACT-Br), a neurological exam and neuro-imaging (MRI) of brain. An extra blood sample will be collected for biomarker studies.

Clinical evaluations include physical exam, vitals, KPS, neurological exam and blood hematology and chemistries (obtained once every month throughout treatment). Neuro-imaging and assessment for response will be performed approximately every 3 months. QOL will be assessed with the KPS rating scale and the FACT-Br questionnaire at screening and then every six months during treatment. Blood will be collected for correlative studies on Day 1 of every even cycle. Any molecular information derived from the correlative studies or clinical care will be associated with the patient's response.

Patients will continue monthly cycles of treatment for 12 cycles or until disease progression or unacceptable toxicity (whichever occurs first). For those in Arm B, patients may continue NovoTTF-200A treatment if temozolomide is discontinued early for toxicity. An end of treatment visit for clinical evaluations and safety assessments will be performed approximately four to six weeks of withdrawing from study treatment. Patients discontinuing study treatment will be followed at months 18 and 24 with tumor assessments if they discontinued from study treatment without disease progression and for survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed low-grade glioma including astrocytoma grade 2, oligodendroglioma grade 2, or oligoastrocytoma grade 2.
* Tumor is supratentorially located and measureable.
* Disease that has not received prior radiation, radiosurgery, chemotherapy, or other investigational treatment directed at the brain tumor at any time. Previous surgical procedures is allowed.
* Age ≥ 18 years.
* Life expectancy > 12 weeks.
* Either not receiving steroids for disease symptoms or are on stable dose of steroids for at least 5 days.
* Karnofsky Performance Status (KPS) ≥ 60%
* Adequate hematologic function evidenced by:

  * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
  * Platelet count ≥ 100 x 109/L
  * Hemoglobin ≥ 9.0 g/dL
* Adequate renal function evidenced by:

  * AST/SGOT and ALT/SPGT ≤ 2.5 X institutional upper limit of normal
  * Total bilirubin ≤ 1.5 x institution's ULN
  * Serum creatinine ≤ 1.5 x institution's ULN

Exclusion Criteria:

* Pilocytic astrocytoma, ganglioglioma, pleomorphic xanthoastrocytoma, or dysembryoplastic neuroepithelial tumors are not eligible.
* Current or anticipated use of other investigational agents.
* Implanted electronic medical device in the brain (e.g., deep brain stimulator, vagus nerve stimulator, programmable shunt).
* Patients who are less than 4 weeks from surgery or have insufficient recovery from surgical-related trauma or wound healing.
* Severe or uncontrolled medical disorder that would, in the investigator's opinion, impair ability to receive study treatment (i.e., uncontrolled diabetes, chronic renal disease, chronic pulmonary disease or active, uncontrolled infection, psychiatric illness/social situations that would limit compliance with study requirements).
* Severe cardiac insufficiency (NYHA III or IV), with uncontrolled and/or unstable cardiac or coronary artery disease.
* Pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
Toxicity associated with treatment with NovoTTF-200A alone and combined with temozolomide | 24 months
  Participants will be assessed for the development of toxicity according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 4.03. Dose adjustments will be made according to the system showing the greatest degree of toxicity.

SECONDARY OUTCOMES:
Efficacy of NovoTTF-200A alone and combined with temozolomide | 24 months
  Participants will be assessed for efficacy of NovoTTF-200A alone and combined with temozolomide as measured by progression free survival (PFS), overall survival (OS), and tumor responses over 24 months.
12-month objective response rate (ORR) of NovoTTF-200A alone and combined with temozolomide | 12 months
  Participants will be assessed for 12-month objective response rate (ORR) of NovoTTF-200A alone and combined with temozolomide in the treatment of adults with newly diagnosed low grade glioma.
Effects of NovoTTF-200A alone and combined with temozolomide on seizure activity | 24 months
  Participants will be assessed for seizure frequency.
Effects of NovoTTF-200A alone and combined with temozolomide on quality of life (QOL) | 24 months
  Participants will be assessed for quality of life using the FACT-Br questionnaire.
Frequency of transformation from low-grade glioma into high-grade glioma | 24 months
  Glioma tumor grade will be assessed over time for transformation to a higher grade.

CONTACTS AND LOCATIONS:
Overall Officials: Santosh Kesari, MD, PhD, Principal Investigator — Saint John's Cancer Institute
Locations (2):
- United States (2):
  - John Wayne Cancer Institute, Santa Monica, California
  - Providence Brain & Spine Institute, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Undecided